CLINICAL TRIAL: NCT00886457
Title: Inhibition of DNA Methylation by 1-hr Infusion of 5-aza-2'-Deoxycytidine (Decitabine) x 10 Days (M-F) With Escalating Doses of Sub-Q Pegylated (PEG) Interferon-alfa 2B (PEG-Intron): A Phase I Study With Molecular Correlates
Brief Title: 5-aza-2-deoxycytidine With Pegylated Interferon-alfa 2B: A Phase I Study With Molecular Correlates
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Nevada Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Schering-Plough (Industry)
Responsible Party: Wolfram Samlowski, MD, Nevada Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVCI-0725; NCI 8224
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Cancer
Keywords: Biopsy proven cancer, which is metastatic or unresectable
MeSH Terms: conditions — Neoplasms | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine plus PEG Interferon-alfa 2B (Experimental): 3.7 mg/m**2 decitabine plus 0, 0.5, 1.5, 3, or 6 mcg/kg PET-Intron
  Interventions: Drug: Decitabine and Pegylated Interferon-Alfa 2B

INTERVENTIONS:
Drug: Decitabine and Pegylated Interferon-Alfa 2B — Patients will receive decitabine 3.7 mg/m2/day i.v. over 1 hour daily in 10 doses over 2 weeks elapsed time (Monday-Friday) every 28 days plus fixed dose of PEG-Intron (0, 0.5, 1.5, 3 or 6 mcg/kg PEG-Intron) weekly by subcutaneous injection in 28-day cycles .

SUMMARY:
The purpose of this study is to assess toxicities of a 1-hr infusion of 5-aza-2'-deoxycytidine (decitabine) x 10 days (M-F) plus escalating doses of weekly subcutaneous PEG-interferon-α (PEG-Intron) in patients with metastatic cancer and to identify the maximum tolerated dose of PEG-Intron in this combination. The pre- and post-treatment samples will be evaluated to identify changes in molecular correlates.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a biopsy proven cancer, which is metastatic or unresectable, for which (in the opinion of the investigator), no curative or more effective treatment exists.
2. Patient must have biopsy accessible tumor and must indicate willingness to undergo biopsies of tumor and normal skin on days 1, 15 and 29.
3. Patient must have measurable disease by RECIST criteria by scans performed within 28 days of study enrollment.
4. Patient may not have untreated brain metastasis. Patients with previously treated brain metastasis must no longer be receiving steroid therapy for the treatment of their brain metastasis.
5. Patient must have a Zubrod performance status of 0 - 2.
6. Prior surgery, radiotherapy or chemotherapy is allowed. The patient must not have received chemotherapy, radiotherapy, surgery, biologic therapy or any other investigational drug for any reason within 28 days prior to registration. Concomitant treatment with other anti-cancer agents or radiotherapy, including investigational agents during the course of study treatment is not allowed.
7. Patients with extensive pelvic irradiation or prolonged nucleoside analogue pretreatment are excluded due to increased risk for hematologic toxicity.
8. Patient must have adequate liver function as defined by a serum bilirubin ≤ 1.5 x the institutional upper limit of normal (IULN), SGOT or SGPT ≤ 2.5 x the institutional upper limit of normal (or ≤ 5 x the institutional upper limit of normal if hepatic metastases is present) obtained within 14 days prior to registration.
9. Patient must have an adequate renal function as defined by a serum creatinine ≤ 1.5 x the institutional upper limit of normal, as well as a calculated or measured creatinine clearance (CrCl) ≥ 50 ml/min.
10. Patient must have an ANC > 1,500/μl, platelet count > 100,000/μl and hemoglobin > 9 gm/dl (this may be achieved by transfusion if needed) obtained within 14 days prior to registration.
11. All patients must be informed of the investigational nature of this study and must provide written acknowledgment of informed consent in accordance with institutional and federal guidelines.
12. Both men and women of all races and ethnic groups are eligible for this trial.
13. Patients must be ≥ 18 years of age.

Exclusion Criteria:

1. Class 3/4 cardiac problems as defined by the New York Heart Association Criteria (e.g., congestive heart failure, myocardial infarction within 2 months of study).
2. Severe and/or uncontrolled concurrent medical disease (e.g., uncontrolled diabetes, uncontrolled chronic renal or liver disease, or active uncontrolled infection, e.g., HIV).
3. Patient must not be pregnant or nursing mothers because PEG-Intron or decitabine may be harmful to the developing fetus and newborn. Women/men of reproductive potential must agree to use an effective contraceptive method. Women of reproductive potential must have a negative serum pregnancy test within 7 days prior to registration. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
4. Medical or psychological conditions that, in the opinion of the investigator, make the patient unable to tolerate or complete the treatment, or to grant reliable informed consent are not eligible for this study.
5. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I, II, or III cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity based on CTCAE Version 3.0 | Daily for 10 days out of 14, and then weekly every 28 days

SECONDARY OUTCOMES:
Genomic DNA methylation and Mage-1 specific promoter methylation in blood cells, tumor and skin | Pretreatment, and then on days 8, 15, 22, and 29

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Samlowski, MD, Principal Investigator — Nevada Cancer Institute
Locations (1):
- Nevada Cancer Institute, Las Vegas, Nevada, United States